CLINICAL TRIAL: NCT02655913
Title: Phase I-II Study of Vitamin C Infusion in Combination With Local mEHT on Non Small Cell Lung Cancer Patients
Brief Title: Safety and Efficacy of Vitamin C Infusion in Combination With Local mEHT to Treat Non Small Cell Lung Cancer
Acronym: VCONSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clifford Hospital, Guangzhou, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHVCONSCLC1842
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer
Keywords: Sodium ascorbate; Non-Small-Cell Lung cancer; Oncothermia; Immune function; Life quality; Tumor marker; Survival time
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ascorbic Acid; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin C+ mEHT+ supportive care (Experimental): Patients will be allocated into 3 Vitamin C infusion dosage groups:
  1g/kg.d,1.2g/kg.d,1.5g/kg.d;3 times a week for 8 weeks(25 infusions);concurrent with Modulated Electro-Hyperthermia (mEHT): 150W x 60 min/session,3 times a week for 8 weeks (25 sessions);together with supportive care.
  Interventions: Drug: vitamin C; Device: Modulated Electro-Hyperthermia (mEHT); Other: Supportive care
- Supportive care (Placebo Comparator): Supportive care focuses on helping patients get relief from symptoms such as nausea, pain, fatigue, or shortness of breath,etc.
  Interventions: Other: Supportive care

INTERVENTIONS:
Drug: vitamin C — Vitamin C infusion, as an alternative anticancer therapy, has been used for many years. In the last 10 years, an increasing number of studies have indicated that VitC in pharmacological concentration can selectively kill cancer cells. Phase I clinical trial showed that VitC(1.5g/kg, 90-120mins, 3 times a week) infusion is safe without significant adverse reactions. A phase II clinical trial indicated that large dose of vitC infusion can reduce toxic side effects from chemo drugs when it was used synergy with chemotherapy.
  Other Names: Sodium Ascorbate
  Arms: vitamin C+ mEHT+ supportive care
Device: Modulated Electro-Hyperthermia (mEHT) — MEHT is a descendant of hyperthermia initially based on nano-thermal but not temperature-dependent effects of electromagnetic fields and special fractal modulation, whose effect could 3-4 times exceed the effect of the overall heating (macroscopic temperature elevation). MEHT does not require hyperthermia-range temperatures and could be performed safely without invasive thermal control. EHY-2000 local machine is used for mEHT in the trial.
  Other Names: Oncothermia
  Arms: vitamin C+ mEHT+ supportive care
Other: Supportive care — Supportive care focuses on helping patients get relief from symptoms such as nausea, pain, fatigue, or shortness of breath,etc.

SUMMARY:
This trial studies efficacy and safety of combination of vitamin C infusion with modulated electro-hyperthermia (mEHT) in treatment of non small cell lung cancer patients.Phase I of this clinical study is to find the tolerable dose and best schedule of the combination of vitamin C infusion and mEHT that can be given to patients with NSCLC. Phase II of this study is to learn if the combination of vitamin C infusion and mEHT can help to control NSCLC and improve quality of life.

DETAILED DESCRIPTION:
Phase I and Phase II clinical trial indicated large dose of vitC infusion is safe and can reduce toxic side effects from chemo drugs when it was used synergy with chemotherapy. The new technology of modulated electro-hyperthermia (mEHT),trade name: oncothermia has been proven efficacy in lung cancer with minimal side effects.The investigators have accumulated some successful cases in the treatment of primary lung cancer by using vitamin C infusion in combination with oncothermia. One diagnosed with squamous cell lung cancer patient survive beyond 5 years only receiving intravenous vitamin C+ mEHT. Based on this, it is necessary to conduct an in-depth study to explore the best treatment protocol for NSCLC patients.

ELIGIBILITY:
Inclusion criteria:

* 18 years old to 70 years
* Primary non small cell lung cancer (stage 3 and 4)
* Subjects must have had their last cancer therapy at least four weeks prior to entry to this study
* The patient must be willing and able to sign the informed consent prior to the start of the trial
* Candidates are not currently receiving cancer therapy (chemotherapy, molecular targeted drug therapy, and radiation therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Willingness to comply with the weekly phone calls between office visits
* Patients must be able to take food orally or have peg tube for feeding
* Life expectancy of at least 6 months

Exclusion Criteria:

* Lung metastasis/not primary non small cell lung cancer
* Glucose-6-phosphate dehydrogenase deficiency (G6PD)
* Vitamin C allergy
* Impossibility to place the patient into the mEHT machine
* Metallic implants or replacements in the treatment area
* Electronic implanted devices anywhere
* Missing or damaged heat-sense nerves or other field-sensitive issues in the treatment area
* Co-morbid conditions that affect survival: end stage congestive heart failure, unstable angina, myocardial infarction (within the past 6 weeks), and uncontrolled blood sugars of greater than 300 mg/dL, known chronic active hepatitis or cirrhosis
* Renal insufficiency as evidenced by serum creatinine of ≥ 1.3mg/dl or evidence of oxalosis by urinalysis
* Chronic hemodialysis
* Iron overload (a ferritin > 500 ng/ml)
* Wilson's disease
* Compromised liver function with evidence of complete biliary obstruction or have a serum bilirubin of 2.0 or liver function tests (AST > 63, ALT > 95) exceeding 1.5 x the upper limit of normal
* Very low white blood cell count (< 1.5 x 10(9)/L), agranulocytosis (< 0.5 x 10(9)/L) or severe anemia
* Pregnant or lactating female
* Current tobacco use
* Evidence of significant psychiatric disorder by history or examination that would prevent completion of the study or preclude informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of vitamin C infusion（1g/kg.d, 1.2g/kg.d,1.5g/kg.d） in combination with oncothermia on NSCLC patients | weekly for up to 8 weeks
  Adverse events, whether volunteered by the study subject, discovered by the investigators during questioning, or detected by physical examination, laboratory tests, or other means will be collected and recorded at each visit. Events will be recorded from the time the consent is signed until 4 weeks after the study protocol is discontinued.

SECONDARY OUTCOMES:
Anti-Tumor Response | 12 weeks after start of treatment
  Tumor markers such as CEA,CYFRA21-1,CA153,SCC will be evaluated at baseline and one month after completion of treatment. Enhanced CT scan will be performed at baseline and one months after completion of treatment to measure the size of the tumor.
Changes in Health Related Quality of Life (EORTC QLQ-C30) | basal,1,2,3,6,12 months follow up
Progression free Survival | CT assessment every 2 months
Overall Survival | every month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Junwen Ou, PhD, Principal Investigator — Clifford Hospital, Guangzhou, China
Locations (1):
- Clifford Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided